CLINICAL TRIAL: NCT02580292
Title: Diagnostic Accuracy of Renal, Carotid, and Aortic Doppler Resistive Indices for Early Diagnosis of Acute Kidney Injury Following Cardiopulmonary Bypass Surgery.
Brief Title: Diagnostic Accuracy of Doppler Resistive Indices for Early Diagnosis of Acute Kidney Injury .
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Milo Engoren, Professor, University of Michigan
Other Study IDs: 1
Record Dates: First submitted 2015-10-17; First posted 2015-10-20 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine if ultrasound measurement of renal and carotid arterial resistive indices are associated with post-cardiac surgery acute kidney injury.

DETAILED DESCRIPTION:
To determine if ultrasound measurement of renal and carotid arterial resistive indices are associated with post-cardiac surgery acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >= 18 years
* undergoing cardiac surgery with cardiopulmonary bypass and transesophageal echocardiography (TEE) probe placement

Exclusion Criteria:

* chronic kidney diseases (estimated GFR < 60 ml/min/1.73m2)
* prior carotid endarterectomy
* known carotid artery stenosis of 50% or greater
* dissection or aneurysm involving renal or carotid arteries
* scheduled aortic or aortic valve surgery
* heart transplant
* intraaortic balloon pump, ventricular assist device, or exctracorporeal membrane oxygenation support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury - Lassnigg grade-minimal | 2nd postoperative day
  Based on change in creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Milo Engoren, Principal Investigator — University of Michigan
Locations (1):
- Cardiovascular Center - University of Michigan, Ann Arbor, Michigan, United States